CLINICAL TRIAL: NCT01483612
Title: "Evaluation of Clinical Outcomes and Costs of a Transferable Interdisciplinary Lifestyle Intervention Pre- and Per-pregnancy in Obese Infertile Women"
Brief Title: Evaluation of Clinical Outcomes and Costs of a Lifestyle Intervention in Obese Infertile Women
Acronym: OF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Principal Investigator, Jean-Patrice Baillargeon, Associate Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIHR/FRN-114125
Record Dates: First submitted 2011-11-25; First posted 2011-12-01 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Female Infertility; Polycystic Ovary Syndrome; Obesity
Keywords: Body Weight; Female; Infertility, Female/therapy; Infertility, Female/physiopathology; Obesity/physiopathology; Polycystic ovary syndrome; Pregnancy; Pregnancy Outcome; Weight Loss
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome; Obesity; Body Weight; Infertility; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Interdisciplinary lifestyle intervention
- control (No Intervention)

INTERVENTIONS:
Behavioral: Interdisciplinary lifestyle intervention — Individual meetings with a dietitian and a kinesiologist at 0, 3, 6 weeks and then every 6 weeks for 18 months or until delivery. A reminder phone call/email will also take place once between each meeting.
  The program also includes 12 group sessions discussing subjects about nutrition, psychology and demonstration of physical activity.
  Other Names: Lifestyle program for obese infertile women
  Arms: Lifestyle counseling

SUMMARY:
BACKGROUND: Obesity increases the risk of polycystic ovary syndrome (PCOS), characterized by anovulatory cycles, but it is also associated with reduced fertility even in ovulatory women. Moreover, obesity increases the costs of assisted human reproduction (AHR) treatments and reduces their efficacy. In addition to fertility disorders, obesity increases significantly the risks of many complications of pregnancy, delivery and neonatal health. However, a modest loss of 5-10% of total body weight can restore ovulation and improve pregnancy rates.

OBJECTIVES: 1) To design and implement a multidisciplinary program for lifestyle management of obese women, or overweight women with PCOS, who seek fertility treatment in a secondary AHR center. 2) To evaluate lifestyle benefits of this program and assess its impact on fertility, pregnancy and neonatal outcomes, as compared to a randomly assigned control group and to similar women seen in tertiary AHR centers. 3) To assess cost per live birth, and other measures of cost-effectiveness, of this program compared to the control group and tertiary AHR centers. 4) To effectively transfer knowledge obtained through these activities to relevant stakeholders in the health care and public health sectors.

METHODS AND APPROACH: In order to design the program for lifestyle management of obesity in infertile women, we will gather a Committee composed of members of our interdisciplinary research team and relevant collaborators. Objectives 2 and 3 - In order to achieve these objectives, 128 obese women (BMI ≥ 30 kg/m²), or overweight women with PCOS (BMI ≥ 27 kg/m²), consulting at the CHUS fertility clinic will be randomized to our lifestyle program, and will suspend fertility treatments for six months, or to standard fertility treatments, which are directly initiated. The results obtained will also be compared to those of women with the same criteria who will consult in 3 tertiary AHR clinics not offering a similar lifestyle management program.

IMPACT: This project is very important as it will generate new knowledge about the implementation, impacts and costs of a new lifestyle management program in obese infertile women. Our project will obtain valuable data on implementability of such a program; on benefits with regard to lifestyle, fertility and maternal and foetal complications during pregnancy; as well as on reduction in cost per live birth and other cost-effectiveness ratio.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI ≥ 30kg/m2) infertile women
* Overweight (BMI ≥ 27kg/m2) infertile women with polycystic ovary syndrome

Exclusion Criteria:

* Women older than 40 years old
* Women who went through bariatric surgery
* Women under IVF
* Women for whome IVF is the only recommended treatment
* Women who do not speak french

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Rates of live birth | Participants who will become pregnant: for the duration before they get pregnant and up to the end of pregnancy, an expected average of 18 months. Participants who will not become pregnant: 18 months

SECONDARY OUTCOMES:
Fertility outcomes | 18 months
Pregnancy outcomes | Participants who will become pregnant: up to the end of pregnancy, an expected average of 18 months of follow-up in the study
Neonatal outcomes | Participants who will become pregnant: up to the end of pregnancy, an expected average of 18 months of follow-up in the study
Clinical outcomes | 18 months
  Evolution of anthropometric measures, change in lifestyle habits, physical fitness level and evolution of readiness for change.
Cost per life birth, and other measures of cost-effectiveness | Participants who will become pregnant: for the duration before they get pregnant and up to the end of pregnancy, an expected average of 18 months. Participants who will not become pregnant: 18 months
  All costs (interventions and complications) to achieve one life birth, including either all women with a life birth or all enrolled women (by intervention arm).
Clinical outcomes in male partners | 18 months
  Evolution of anthropometric measures and change in lifestyle habits in male partners.
Clinical outcomes of female participants | 18 months
  Evolution of anthropometric measures, changes in lifestyle habits (diet, exercise, alcohol, tobacco), physical fitness level, evolution of readiness for change, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Patrice Baillargeon, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] St-Laurent A, Belan M, Jean-Denis F, Langlois MF, Pesant MH, Carranza-Mamane B, Duval K, Morisset AS, Baillargeon JP. An interdisciplinary intervention improves lifestyle behaviours in women living with obesity and subfertility: A secondary analysis of a randomized controlled trial. Clin Nutr ESPEN. 2025 Aug;68:457-464. doi: 10.1016/j.clnesp.2025.05.036. Epub 2025 May 28. PMID 40447224
- [Derived] Duval K, Langlois MF, Carranza-Mamane B, Pesant MH, Hivert MF, Poder TG, Lavoie HB, Ainmelk Y, St-Cyr Tribble D, Laredo S, Greenblatt E, Sagle M, Waddell G, Belisle S, Riverin D, Jean-Denis F, Belan M, Baillargeon JP. The Obesity-Fertility Protocol: a randomized controlled trial assessing clinical outcomes and costs of a transferable interdisciplinary lifestyle intervention, before and during pregnancy, in obese infertile women. BMC Obes. 2015 Dec 1;2:47. doi: 10.1186/s40608-015-0077-x. eCollection 2015. PMID 26635965